CLINICAL TRIAL: NCT03509337
Title: Changes in the Tension of the Flexor Carpi Ulnar Muscle With the Tensioning of the Ulnar Nerve by Shear-wave Elastography: a Pilot Study
Brief Title: Changes in the Ulnar Tissues by Shear-wave Elastography
Status: Completed | Type: Observational
Sponsor: Guadarrama Hospital (Other)
Collaborators: Universidad Francisco de Vitoria (Other)
Responsible Party: Principal Investigator, J. Nicolas Cuenca Zaldivar, Rehabilitation Service Principal Investigator, Guadarrama Hospital
Other Study IDs: 3.0
Record Dates: First submitted 2018-04-17; First posted 2018-04-26 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Elastography; Soft Tissue; Muscle Tonus
Keywords: Elastography, Nervous tissue, Muscle tonus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: shear-wave elastography — Measurement by shear-wave elastography of the nerve, muscle and ulnar tendon before and after the tension of the ulnar nerve

SUMMARY:
A single-center, observational, prospective, single cohort study with before-after design. Evaluation by shear-wave elastography, measured in kilopascals (KPa), of the muscle, tendon and cubital nerve, before and after the maneuver of putting in tension of the ulnar nerve.

DETAILED DESCRIPTION:
Once each subject has signed the informed consent document and it has been verified that the inclusion criteria are met, it will be assigned the same identification number (ID) that is related to its Clinical History (CH) by simple coding; custody of the file with the relationship of each ID with its CH will be the responsibility of the principal investigator.

Body placement: The participants will be placed in the supine position with the hips and knees bent, in such a way that the soles of the feet rest on the plane of the stretcher. the palm of the hand of the left extremity will rest on the abdomen and the head in a neutral position, with the maximum relaxation of the sternocleidomastoids.

Upper limb placement: The right extremity will be placed in abduction of 90°, the elbow to flexion of 10° and the forearm to 30° of supination. Wrist and joints metacarpophalangic (mcf), proximal interphalangeal (ifp) and distal interphalangeal (ifp) of the first three fingers in full extension. The articulations mcf, ifp, ifd of the fourth and fifth fingers in a relaxed position. In this position, the first ultrasound measurement will be taken.

Tension maneuver of the ulnar nerve: An expert researcher in mobilization of neural tissue will perform an extension of fourth and fifth finger, respecting the initial parameters that are maintained in position by the splint. To do this, he will use the index and middle of his left hand and make a contact on the palmar side of the fingers and a back pressure with the thumb on the back of the hand. Next, it will extend the fingers until the exponential resistance following the path of elastic deformation (linear resistance) of the tensioned tissues is perceived. At this time the new ultrasound record will be made.

Ultrasound records: A Toshiba ai800 ultrasound scanner (Toshiba Medical Corporation, Japan) with a multifrequency linear probe plt-1005bt 14l5 (5-14 Mhz) will be used. The identification number (ID) registered in the ultrasound will correspond to the participant number.

The same researcher, with experience in the acquisition and management of medical images, will perform the ultrasound and in-line measurements of the images obtained.

The ultrasound will be obtained in a pre and post-median situation after the neural tension put on by the expert investigator in manual therapy and a label will be consigned in the images indicating if the acquisition was "pre" or "post".

To perform the acquisition of the images the probe wil be positioned on the skin of the forearm with minimal pressure and with angulation such that there is no anisotropy. The anatomical region where the myotendinous junction of the flexor carpi ulnaris muscle and the ulnar nerve is observed will be searched transversally. the parameters of emission power, general gain, depth of the image, position of the focus and frequency of emission will be adapted to obtain a quality image. The protocol will be the following:

* 2d image in transverse plane.
* 2d image in longitudinal plane.
* Shear-wave elastography in longitudinal plane.
* Measurement of the images: They will be carried out off-line using the elastography software of the team itself once all the participants have been explored. three regions of interest (ROIs) adjacent to each other will be established in the body of the ulnar nerve, three in the distal area of the flexor carpi ulnaris muscle and three in the tendinous body of the same muscle. The size of the ROI should include the entire body of the mentioned structures.
* The average value of the three ROIs will be written down in units of pressure (KPa).

ELIGIBILITY:
Inclusion Criteria:

* Francisco de Vitoria University student.
* Age between 18 and 26 years old.

Exclusion Criteria:

* History of neuropathies in upper limbs.
* Slight neck pain in the last 6 months of traumatic origin.
* Neck pain in the last 3 months.
* episodes of moderate / severe neck pain in the last year.
* History of fracture or dislocation in the upper extremity.
* Surgical history in the upper extremity.
* Cervical symptomatology or upper limb at the present time.

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers recruited among the students of the Francisco de Vitoria University.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
elastographic soft tissue tension (KPa) | 1 day
  Tension (KPa) in the nerve, muscle and ulnar tendon measured by elastography shear-wave before and after putting the ulnar nerve in tension

CONTACTS AND LOCATIONS:
Overall Officials: J. Nicolas Cuenca Zaldivar, Principal Investigator — Guadarrama Hospital
Locations (1):
- J.Nicolas Cuenca Zaldivar, Guadarrama, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
The statistical analysis plan and the analytical code will be available in .html and .rmd format as well as the file with the raw data.
Supporting Information: SAP, Analytic Code
Time Frame: The data will be available permanently once the statistical analysis is complete.
Access Criteria: The data will be available freely and publicly.
URL: https://github.com/jcuenzal/Changes-in-the-tension-of-the-flexor-carpi-ulnar-muscle-with-the-tensioning-of-the-ulnar-nerve-by-sh.git